CLINICAL TRIAL: NCT06361173
Title: Spanish BMT4me Usability & Acceptability
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Micah Skeens, Principal Investigator, Nationwide Children's Hospital
Other Study IDs: STUDY00004127
Record Dates: First submitted 2024-04-02; First posted 2024-04-11 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Bone Marrow Transplant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spanish-speaking caregivers: Spanish-speaking caregivers recruited from Nationwide Children's Hospital and Columbia University Irving Medical Center to pilot test a Spanish a transcreated version of the BMT4me app
  Interventions: Other: BMT4me

INTERVENTIONS:
Other: BMT4me — Caregivers will pilot test a Spanish version of the BMT4me app at a single time point.

SUMMARY:
The objective of this project is to trans-create, conduct user testing of a previously developed and piloted mHealth app, and user acceptability with parents of children in the acute phase post-allogeneic hematopoietic stem cell transplant (HSCT). Nationwide Children's Hospital (NCH) will be the primary data collection site and Columbia University Irving Medical Center will be a secondary site.

ELIGIBILITY:
Inclusion Criteria:

Eligible caregivers must have children who:

1. Are 0-17 years old
2. Underwent HCT
3. Are planned for discharge prior to day 100 post-transplant

Primary caregivers must:

1. Be Spanish speaking
2. Be ≥18 years old
3. Have a smartphone (iOS or Android) capable of downloading apps

Exclusion Criteria:

(a) Children or caregivers with pre-existing neurodevelopmental disorder/disability or a pervasive developmental disorder will be excluded from this study.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will recruit 30 self-identified Spanish speaking primary caregivers of children post-HCT at two institutions.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Assess app usability using the System Usability Scale (SUS) | 6/1/24 - 5/1/26
  Data collected using the System Usability Scale (SUS) will provide insight to the usability of the Spanish BMT4Me app in its current form. he SUS is a 10-item questionnaire routinely used to evaluate the functionality and acceptability of mHealth apps. The SUS is scored on a scale, giving a score from from 0 to 100 where 100 is considered the highest rating of usability. A score of > 68 is considered above average.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be shared upon request.